CLINICAL TRIAL: NCT03969056
Title: Applying Artificial Intelligence to a Physical Activity Intervention in Patients With Elevated Blood Pressure- a Pilot Randomized Controlled Trial
Brief Title: AI Activity Study in Patients With Elevated Blood Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-26452
Record Dates: First submitted 2019-05-20; First posted 2019-05-31 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Artificial Intelligence; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence (AI) Activity group (Experimental): Participants in this group receive an AI based intervention (automated and personalized daily step goal intervention involving a sophisticated activity analytics algorithm using advanced statistics and machine learning and message)
  Interventions: Behavioral: Artificial Intelligence (AI) Activity
- Control group (Active Comparator): Participants in this group receive a standardized and fixed 10,000 daily steps goal intervention.
  Interventions: Behavioral: 10,000 steps

INTERVENTIONS:
Behavioral: Artificial Intelligence (AI) Activity — The intervention provides participants with an automated and personalized daily step goal intervention involving a sophisticated activity analytics algorithm using advanced statistics and machine learning.
  Arms: Artificial Intelligence (AI) Activity group
Behavioral: 10,000 steps — The intervention provides participants with an automated daily 10,000 step goal intervention
  Arms: Control group

SUMMARY:
In this pilot RCT, a total of 40 adults with hypertension will be randomized to either an artificial intelligence (AI) physical activity intervention group or an active control group with a 1 to 1 ratio after completing a 2-week run-in period and 4-week training. The AI intervention group will receive an automated and personalized daily step goal intervention involving a sophisticated activity analytics algorithm using advanced statistics and machine learning, while the active control group will receive a standardized and fixed 10,000 daily steps goal. Both groups will receive an identical smartphone app (app content differs between the two groups) and ActiGraph GT9X Link to assess objectively measured physical activity (primary outcome) during the study period.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* systolic blood pressure between 130 mmHg to 180 mmHg or/and diastolic blood *pressure between 80 to 100 mmHg in a research office
* speaking and reading English
* being physically inactive at work or during leisure time and willing to be physically active
* having an iPhone 8 or newer or an Android Lollipop or newer

Exclusion Criteria:

* self-reported diagnosis of coronary heart disease, medical condition or other physical problem necessitating special attention in an exercise program (e.g., cancer, eating disorder, uncontrolled diabetes)
* current participation in a lifestyle modification program or research study
* self-report of being currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in weekly daily average steps | Baseline (run-in period), 4 week-test period, and 3-month intervention period
  measured by ActiGraph GT9X Link]
Duration (minutes) of moderate to vigorous intensity physical activity (MVPA) per day | Baseline (run-in period), 4 week-test period, and 3-month intervention period
  measured by ActiGraph GT9X Link]

SECONDARY OUTCOMES:
Changes in Systolic blood pressure (SBP) | Baseline (run-in period), 4 week-test period, and 3-month intervention period
Changes in diastolic blood pressure (DBP) | Baseline (run-in period), 4 week-test period, and 3-month intervention period
aortic stiffness | Baseline (run-in period), 4 week-test period, and 3-month intervention period
  measured by SphigmoCor XCEL system
sodium intake | Baseline (run-in period), 4 week-test period, and 3-month intervention period
  as measured in 24-hour urine samples
Changes in weight | Baseline (run-in period), 4 week-test period, and 3-month intervention period
Changes in Body Mass Index (BMI) | Baseline (run-in period), 4 week-test period, and 3-month intervention period
  using weight and height to calculate

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimi Fukuoka, PhD, RN, FAAN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No